CLINICAL TRIAL: NCT03221270
Title: Targeting Auditory Hallucinations With Alternating Current Stimulation
Acronym: STILL3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-1364; 4R33MH105574-03 (NIH)
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Results first posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-01

CONDITIONS: Schizophrenia; Schizo Affective Disorder
Keywords: tACS; Sham; Auditory Hallucinations; Schizophrenia; Schizo Affective Disorder; EEG
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Hallucinations

STUDY DESIGN:
Intervention Model Description: Participants will initially be randomized to either sham or 10 Hz tACS for the 5 consecutive days of stimulation. Participants will then be re-randomized to either sham or 10 Hz tACS for the 8 weeks of maintenance stimulation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double blind, randomized clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- tACS Treatment & tACS Maintenance (Experimental): 10 Hz (alpha) tACS with a peak-to-peak amplitude of 2 mA for 20 minutes twice daily during 5 consecutive days of stimulation. 10 Hz (alpha) tACS with a peak-to-peak amplitude of 2 mA for 40 minutes once weekly for 8 weeks of maintenance stimulation.
  Interventions: Device: tACS treatment week; Device: Maintenance tACS
- Sham tACS Treatment & Sham tACS Maintenance (Sham Comparator): 10 seconds of ramp in to 1 minute of 10 Hz (alpha) tACS with a ramp out of 10 seconds for a total of 80 seconds of stimulation twice daily during 5 consecutive days of stimulation. 10 seconds of ramp in to 1 minute of 10 Hz (alpha) tACS with a ramp out of 10 seconds for a total of 80 seconds of stimulation once weekly for 8 weeks of maintenance stimulation.
  Interventions: Device: tACS sham week; Device: Maintenance Sham tACS
- Sham tACS Treatment & tACS Maintenance (Other): 10 Hz (alpha) tACS with a peak-to-peak amplitude of 2 mA for 40 minutes once weekly for 8 weeks of maintenance stimulation.10 Hz (alpha) tACS with a peak-to-peak amplitude of 2 mA for 40 minutes once weekly for 8 weeks of maintenance stimulation.
  Interventions: Device: tACS sham week; Device: Maintenance tACS
- tACS Treatment & Sham tACS Maintenance (Other): 10 Hz (alpha) tACS with a peak-to-peak amplitude of 2 mA for 20 minutes twice daily during 5 consecutive days of stimulation. 10 seconds of ramp in to 1 minute of 10 Hz (alpha) tACS with a ramp out of 10 seconds for a total of 80 seconds of stimulation once weekly for 8 weeks of maintenance stimulation.
  Interventions: Device: tACS treatment week; Device: Maintenance Sham tACS

INTERVENTIONS:
Device: tACS treatment week — 10 Hz sine wave stimulation with a peak-to-peak amplitude of 2 mA for 20 minutes twice for 5 consecutive days.
  Other Names: Neuroconn DC Stimulator
  Arms: tACS Treatment & Sham tACS Maintenance; tACS Treatment & tACS Maintenance
Device: tACS sham week — 10Hz sine wave stimulation with a peak-to-peak amplitude of 2 mA for 10 seconds twice a day for 5 consecutive days.
  Other Names: Neuroconn DC Stimulator
  Arms: Sham tACS Treatment & Sham tACS Maintenance; Sham tACS Treatment & tACS Maintenance
Device: Maintenance tACS — 10 Hz sine wave stimulation with a peak-to-peak amplitude of 2 mA for 40 minutes once a weekly for 8 weeks.
  Other Names: Neuroconn DC Stimulator
  Arms: Sham tACS Treatment & tACS Maintenance; tACS Treatment & tACS Maintenance
Device: Maintenance Sham tACS — 10Hz sine wave stimulation with a peak-to-peak amplitude of 2 mA for 10 seconds once a week for 8 weeks.
  Other Names: Neuroconn DC Stimulator
  Arms: Sham tACS Treatment & Sham tACS Maintenance; tACS Treatment & Sham tACS Maintenance

SUMMARY:
Investigating the effects of non-invasive transcranial alternating current stimulation (tACS) as a treatment for auditory hallucinations in patients with schizophrenia.

DETAILED DESCRIPTION:
The investigator's primary objective is to provide further evidence for the effectiveness of transcranial alternating current stimulation (tACS) to treat auditory hallucinations and to collect preliminary data on whether maintenance stimulation sessions can prolong the duration of stimulation-induced clinical benefits. The investigators will be looking into effects of tACS to re-normalize pathological alpha oscillations in the dorso-lateral prefrontal cortex (dl-PFC) of patients with schizophrenia or schizo-affective disorder by comparing Auditory Hallucination Rating Scale (AHRS) scores immediately before the first stimulation session, immediately after the last stimulation session, and at the end of the 8 weeks of maintenance sessions. As a secondary objective, the investigators will assess the differential clinical effects of active sham and 10Hz tACS on electroencephalogram (EEG) measures of alpha oscillations. The investigators will also be using source localization techniques in EEG analysis, based on individual locations of the scalp electrodes and anatomical structures with the use of structural magnetic resonance imaging (sMRI).

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia, any subtype, or schizoaffective disorder with refractory hallucinations. Duration of illness >1 year
* 18 - 70 years old
* Clinical stable for at least 12 weeks i.e. not requiring any hospitalization or a change in level of care
* On current antipsychotic doses for at least 4 weeks
* Experience at least 3 auditory hallucinations per week
* Stable auditory hallucinations as demonstrated by having less than or equal to 20% change in AHRS scores across a 2 week interval during the screening period
* Capacity to understand all relevant risks and potential benefits of the study and to provide written informed consent, OR has a legal guardian who can provide the informed consent on the patient's behalf with the patient providing written assent to participate

Exclusion Criteria:

* DSM-IV diagnosis of alcohol or substance abuse (other than nicotine) within the last month or a DSM-IV diagnosis of alcohol or substance dependence (other than nicotine) within the last 6 months
* Positive urine test of cannabis, cocaine, amphetamine, barbiturates, opiates
* Current treatment (within 4 weeks) with psychotropic agents including benzodiazepines that are taken on a daily basis (limit prn use to greater than 48 hours before participating in a study session)
* Medical or neurological illness (unstable cardiac disease, AIDS, malignancy, liver or renal impairment) or treatment for a medical disorder that could interfere with study participation
* history of traumatic brain injury that required subsequent cognitive rehabilitation, or caused cognitive sequelae
* A difference of greater than 20% in AHRS scores between screening visits
* Prior brain surgery
* Any brain devices/implants, including cochlear implants and aneurysm clips
* Co-morbid neurological condition (e.g. seizure disorder, brain tumor)
* Non English speakers
* Female participants who are pregnant, nursing, or unwilling to use appropriate birth control measures during study participation
* Anything that, in the opinion of the investigator, would place the participant at increased risk or preclude the participants' full compliance with or completion of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — University of North Carolina at Chapel Hill - Department of Psychiatry
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Brunelin J, Mondino M, Gassab L, Haesebaert F, Gaha L, Suaud-Chagny MF, Saoud M, Mechri A, Poulet E. Examining transcranial direct-current stimulation (tDCS) as a treatment for hallucinations in schizophrenia. Am J Psychiatry. 2012 Jul;169(7):719-24. doi: 10.1176/appi.ajp.2012.11071091. PMID 22581236
- [Background] Frohlich F, Burrello TN, Mellin JM, Cordle AL, Lustenberger CM, Gilmore JH, Jarskog LF. Exploratory study of once-daily transcranial direct current stimulation (tDCS) as a treatment for auditory hallucinations in schizophrenia. Eur Psychiatry. 2016 Mar;33:54-60. doi: 10.1016/j.eurpsy.2015.11.005. Epub 2016 Feb 8. PMID 26866874

RESULTS

PARTICIPANT FLOW:
Groups:
- tACS Treatment & tACS Maintenance: 10 Hz (alpha) transcranial alternating current stimulation (tACS) with a peak-to-peak amplitude of 2 mA for 20 minutes twice daily during 5 consecutive days of stimulation. 10 Hz (alpha) tACS with a peak-to-peak amplitude of 2 mA for 40 minutes once weekly for 8 weeks of maintenance stimulation.
  tACS treatment week: 10 Hz sine wave stimulation with a peak-to-peak amplitude of 2 mA for 20 minutes twice for 5 consecutive days.
  Maintenance tACS: 10 Hz sine wave stimulation with a peak-to-peak amplitude of 2 mA for 40 minutes once a weekly for 8 weeks.
- Sham tACS Treatment & tACS Maintenance: 10 seconds of ramp in to 1 minute of 10 Hz (alpha) tACS with a ramp out of 10 seconds for a total of 80 seconds of stimulation twice daily during 5 consecutive days of stimulation. 10 Hz (alpha) tACS with a peak-to-peak amplitude of 2 mA for 40 minutes once weekly for 8 weeks of maintenance stimulation.
  tACS sham week: 10Hz sine wave stimulation with a peak-to-peak amplitude of 2 mA for 10 seconds twice a day for 5 consecutive days.
  Maintenance tACS: 10 Hz sine wave stimulation with a peak-to-peak amplitude of 2 mA for 40 minutes once a weekly for 8 weeks.
Period: Overall Study
Arm/Group | tACS Treatment & tACS Maintenance | Sham tACS Treatment & Sham tACS Maintenance | Sham tACS Treatment & tACS Maintenance | tACS Treatment & Sham tACS Maintenance
Started | 8 | 6 | 5 | 6
Completed 5-Day Treatment | 8 | 6 | 5 | 6
Completed 8-Week Maintenance | 4 | 6 | 5 | 5
Completed | 4 | 6 | 5 | 5
Not Completed | 4 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | tACS Treatment & tACS Maintenance | Sham tACS Treatment & Sham tACS Maintenance | Sham tACS Treatment & tACS Maintenance | tACS Treatment & Sham tACS Maintenance | Total
Number analyzed (Participants) | 8 | 6 | 5 | 6 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (12.5) | 45.0 (9.6) | 34.2 (10.1) | 40.4 (11.7) | 39.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 2 | 9
  Male | 5 | 4 | 3 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 5 | 6 | 4 | 5 | 20
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 4 | 3 | 12
  White | 4 | 3 | 0 | 2 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 6 | 5 | 6 | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean Auditory Hallucination Rating Scale (AHRS) Score
Description: The Auditory Hallucination Rating Scale (AHRS) measures the severity of auditory hallucinations in the past week. The scale assess frequency, duration, location, loudness, belief of origin of voices, negative content, distress, disruption to life, and control over voices. All items are measured on a scale of 0 to 4, with a total possible score of 44. Higher scores indicate higher severity of auditory hallucinations.
Time Frame: Baseline, immediately after five days of stimulation, and immediately after the 8th week of maintenance stimulation.
Population: Data for missing sessions was carried forward by replacing with the most recently completed session values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tACS Treatment & tACS Maintenance | Sham tACS Treatment & Sham tACS Maintenance | Sham tACS Treatment & tACS Maintenance | tACS Treatment & Sham tACS Maintenance
Number analyzed (Participants) | 8 | 6 | 5 | 6
score on a scale
  Baseline (T1) | 25.00 (7.37) | 23.17 (7.03) | 23.40 (6.54) | 19.00 (6.75)
  End of 5-Day Treatment Week | 25.13 (8.01) | 21.00 (5.93) | 25.60 (6.84) | 19.83 (5.08)
  End of Maintenance | 23.94 (9.63) | 17.58 (7.10) | 26.40 (6.82) | 15.67 (4.97)
Statistical Analysis 1: Comparison: tACS Treatment & tACS Maintenance vs Sham tACS Treatment & Sham tACS Maintenance vs Sham tACS Treatment & tACS Maintenance vs tACS Treatment & Sham tACS Maintenance; Test type: Superiority — alternative hypothesis: true difference in means is greater than 0; p = 0.66, t-test, 1 sided; Median Difference (Final Values) = -0.43, 95% CI 1-sided [lower limit -2.25]

2. Secondary Outcome: Percentage of Signal Change in the Average Alpha Oscillation Power From Eyes-Open Resting State Electroencephalogram (EEG)
Description: Eyes-open but at rest EEG data was sampled using a 128-channel Geodesic EEG system. Alpha power spectral density was estimated using the Welch's method (in 2s Hamming windows with 0.5s overlap and 0.1 Hz spectral resolution). Aperiodic components were removed before extracting the individual alpha frequency (IAF; peak with the highest power density between 7 to 12 Hz, with consistent presence during the eyes-open blocks across all sessions). All spectra were visually inspected to confirm IAF choice. We computed the percent signal change of alpha power for each session relative to the baseline session:% change_n=(P_baseline-P_n)/P_baseline where P_n is the alpha power in the n-th session, and P_baseline is the alpha power in the baseline session.
Time Frame: Change from baseline to immediately after five days of stimulation, and immediately after the 8th week of maintenance stimulation.
Population: Data for missing sessions was carried forward by replacing with the most recently completed session values.
Measure: Mean (Standard Deviation); unit: percentage of signal change
Arm/Group | tACS Treatment & tACS Maintenance | Sham tACS Treatment & Sham tACS Maintenance | Sham tACS Treatment & tACS Maintenance | tACS Treatment & Sham tACS Maintenance
Number analyzed (Participants) | 8 | 6 | 5 | 6
percentage of signal change
  Average alpha power change from baseline to after 5 days of consecutive stimulation. | 1.64 (22.77) | 4.48 (41.82) | -11.64 (21.00) | 18.62 (35.98)
  Average alpha power change from baseline to after the final stimulation session at week 8. | 31.35 (57.06) | 4.40 (24.94) | -22.21 (14.70) | 40.96 (50.40)

3. Secondary Outcome: Average Score on the Positive and Negative Syndrome Scales (PANSS)
Description: The Positive and Negative Syndrome Scale (PANSS) is a 30-item clinician-administered scale. Each item is scored on a seven point scale, representing increasing levels of psychopathology (1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme). Each item is rated in consultation with the definitions and criteria provided in the manual. Seven items constitute the positive scale, seven items make up the negative scale, and the remaining sixteen make up a general psychopathology scale. Therefore, the potential ranges are 7 to 49 for both positive and negative scales, and 16 to 112 for the General Psychopathology Scale.
Time Frame: Baseline, immediately after five days of stimulation, and immediately after the 8th week of maintenance stimulation.
Population: Data for missing sessions was carried forward by replacing with the most recently completed session values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tACS Treatment & tACS Maintenance | Sham tACS Treatment & Sham tACS Maintenance | Sham tACS Treatment & tACS Maintenance | tACS Treatment & Sham tACS Maintenance
Number analyzed (Participants) | 8 | 6 | 5 | 6
score on a scale
  Mean Positive Symptoms Scale at Baseline | 19.5 (4.4) | 16.8 (5.4) | 18.0 (2.7) | 19.0 (6.8)
  Mean Negative Symptoms Scale at Baseline | 16.1 (6.3) | 18.2 (5.3) | 16.8 (4.2) | 13.8 (5.7)
  Mean General Psychopathology Symptoms Scale at Baseline | 36.5 (11.5) | 31.0 (11.6) | 33.0 (5.0) | 27.7 (7.1)
  Mean Positive Symptoms Scale after 5 days of stimulation | 18.6 (4.0) | 17.3 (5.2) | 16.6 (3.4) | 17.2 (4.7)
  Mean Negative Symptoms Scale after 5 days of stimulation | 15.5 (5.1) | 17.7 (3.5) | 17.6 (6.5) | 15.0 (7.0)
  Mean General Psychopathology Symptoms Scale after 5 days of stimulation | 32.0 (8.4) | 29.7 (10.3) | 22.6 (2.4) | 26.0 (5.7)
  Mean Positive Symptoms Scale after 8 weeks of stimulation | 18.3 (3.9) | 15.7 (5.2) | 17.2 (2.17) | 17.0 (3.2)
  Mean Negative Symptoms Scale after 8 weeks of stimulation | 16.3 (5.3) | 15.5 (5.0) | 16.8 (4.4) | 15.7 (6.8)
  Mean General Psychopathology Symptoms Scale after 8 weeks of stimulation | 32.5 (5.8) | 28.8 (11.0) | 31.20 (2.5) | 25.3 (5.4)

4. Secondary Outcome: Brief Assessment Cognition in Schizophrenia (BACS)
Description: The Brief Assessment of Cognition in Schizophrenia (BACS) is a clinically administered pen- and -paper battery of neurocognitive tests. The tasks administered in person included verbal memory, digit sequencing, token motor task, semantic fluency, letter fluency, symbol coding, and the tower of London task. The scores on each subtest were not normalized or scaled, values from each test were summed. In this sample the total summed scores ranged 112-296 with a standard deviation of 39.61. Higher values represent greater cognitive performance.
Time Frame: Baseline, immediately after five days of stimulation, and immediately after the 8th week of maintenance stimulation.
Population: Data for missing sessions was carried forward by replacing with the most recently completed session values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tACS Treatment & tACS Maintenance | Sham tACS Treatment & Sham tACS Maintenance | Sham tACS Treatment & tACS Maintenance | tACS Treatment & Sham tACS Maintenance
Number analyzed (Participants) | 8 | 6 | 5 | 6
units on a scale
  Mean BACS at Baseline | 194.63 (34.45) | 184.00 (31.82) | 220.40 (39.51) | 215.00 (25.91)
  Mean BACS after five days of stimulation | 208.38 (44.75) | 188.17 (22.14) | 243.20 (45.10) | 208.33 (48.70)
  Mean BACS after 8 weeks of stimulation | 210.00 (52.21) | 194.83 (24.20) | 235.40 (49.20) | 220.17 (30.93)

5. Other Pre Specified Outcome: Electroencephalogram (EEG) Auditory Task
Description: The investigators will compare alpha oscillation power from resting state EEG recordings on the first and last day of stimulation. The investigators will also collect EEG recordings data at the 1st, 3rd, and final maintenance stimulation visits.
Time Frame: Change across time from baseline measurement to final maintenance stimulation
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Auditory Hallucination Rating Scale (AHRS)
Description: The investigators will compare the AHRS scores from baseline across the 8 weeks of maintenance stimulation sessions as an outcome measure.
Time Frame: Change from Baseline AHRS at final maintenance stimulation session.
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: The investigators will compare the PANSS scores from baseline across the 8 weeks of maintenance stimulation sessions as an outcome measure.
Time Frame: Change from Baseline PANSS at final maintenance stimulation session.
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Brief Assessment Cognition in Schizophrenia (BACS)
Description: The investigators will compare the BACS scores from baseline across the 8 weeks of maintenance stimulation sessions as an outcome measure.
Time Frame: Change from Baseline BACS at final maintenance stimulation session.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at each visit during the 5-day treatment and the 8-week maintenance over an approximate 9-week period using a stimulation side effects questionnaire provided to participants after every presentation of each intervention. Data were not collected beyond the eighth maintenance treatment week.
Arm/Group | tACS Treatment & tACS Maintenance | Sham tACS Treatment & Sham tACS Maintenance | Sham tACS Treatment & tACS Maintenance | tACS Treatment & Sham tACS Maintenance
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 3/8 | 0/6 | 1/5 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | tACS Treatment & tACS Maintenance (N=8) | Sham tACS Treatment & Sham tACS Maintenance (N=6) | Sham tACS Treatment & tACS Maintenance (N=5) | tACS Treatment & Sham tACS Maintenance (N=6)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burning Sensation on Scalp (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscular Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT03221270/Prot_SAP_000.pdf